CLINICAL TRIAL: NCT00711945
Title: Growth Relapse and Outcomes With Therapy 1:Factors Determining Poor Outcomes in Pediatric Crohn"s Disease
Brief Title: Growth Relapse and Outcomes With Therapy 1
Acronym: GROWTH1
Status: Completed | Type: Observational
Sponsor: European Society of Pediatric Gastroenterology, Hepatology and Nutrition (Other)
Responsible Party: Principal Investigator, Arie Levine MD, Director, Wolfson Medical Center
Other Study IDs: GROWTH1
Record Dates: First submitted 2008-07-07; First posted 2008-07-09 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: Crohn's Disease; Pediatric Onset
Keywords: Crohn's disease; Relapse; outcomes; growth
MeSH Terms: conditions — Crohn Disease; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum for antiglycan antibodies stool for calprotectin
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Pediatric Crohn's Disease is a life long disease , presenting early in life.As such , it is imperative to be able to evaluate the risk for more severe disease and poorer outcomes when making the decision which therapies to offer our patients. These decisions should be based according to longer-term disease outcomes, such as whether they prevent disease relapse or prolong remission [10-12]. However, for the most part, previous studies were not designed to yield predictive parameters that could allow a clinician to differentiate which patients are at a higher risk for relapse, or more likely to to have serious attacks or complications of the disease or therapy. The ability to predict these risks would impact dramatically the way CD patients are treated, allowing the clinician to tailor therapy, both type and intensity, to each patient's individual risk for relapse and outcomes.In the present first phase of the study , we will attempt to identify factors that predict relapse of the disease, focusing on the use of calprotectin at onset and after clinical remission, and on the use of anti-glycan antibodies, as well as disease severity, site and phenotype.

DETAILED DESCRIPTION:
This proposal describes the first prospective large pediatric cohort study designed to look simultaneously, from disease onset, at clinical, inflammatory, serological and therapeutic parameters of CD, with standardized treatment regimens and long-term follow-up. The exploratory study will delineate whether a sub-clinical inflammatory parameter (calprotectin), performed post-treatment and after achieving remission, is indeed predictive of time to relapse or relapse rate. We anticipate that patients with low calprotectin levels are significantly less likely to relapse during the follow-up period, while patients with persistent inflammation after induction of remission (high calprotectin levels) are more likely to relapse early. We will also evaluate the relationships between various clinical and sub-clinical parameters and CD disease outcomes, as well as the influence of treatments on these parameters. Greater knowledge about the relationship between inflammatory and serological markers, treatments chosen, and CD outcome will improve disease control in the clinic and may offer insights as to how the clinician can modify the course of CD. Furthermore, this study should answer the following question: in patients with clinical improvement but ongoing inflammation, should we treat according to clinical symptoms or should we treat according to sub-clinical laboratory data? Finally, without industry bias, this study may offer ultimately the ability to model factors predictive of poorer outcomes, and to compare the long-term benefits or hazards of treatments in use today.

The framework of the proposed study is development prospectively of an incident cohort of ~300 +/- 30 newly diagnosed cases of CD over a period of two years by a team of pediatric gastroenterologists that represent approximately 20 European IBD centers (the ESPGHAN 'Porto' group). Multiple clinical and laboratory parameters will be recorded serially at intervals in a standardized, pre-agreed format, at initial presentation and for the subsequent 18 months.

At initial presentation, each IBD clinic will confirm independently diagnosis of CD, as opposed to any other inflammatory bowel condition, according to the Porto criteria . These newly diagnosed untreated pediatric patients with CD must be under the age of 18. Exclusion criteria will include abdominal surgery, pregnancy and indeterminate colitis. All participating centers will file an IRB within their own organization. Consent will be sought from each patient or patient's guardian and documented in their native language. Participation in this study does not entail any novel therapeutic intervention, and as such does not pose any risk to the patient. Most of the data to be collected during the study are collected routinely during care of a CD pediatric patient, although there will be extra blood and stool samples taken. Since it is standard to take blood for other tests during these visits, for example to assess disease activity or the presence of anemia or other complications, it is not anticipated that the blood draws will inhibit participation. Therefore, we predict that almost all eligible patients (80%) that present at 'Porto' group centers will be enrolled in this study. At each visit, a clinician will evaluate and record the location of disease, height and weight, as well as disease activity (Pediatric Crohn's Disease Activity Index, PCDAI; and CRP . A stool sample will be taken at all visits for assessing fecal calprotectin (a measure of intestinal inflammation . Any disease complications, such as fistulae, abscess or strictures will also be noted as well as the type (if any) of treatment to be administered. There will be 6 predetermined standard visits at 0, 8, 12, 26, 52 and 78 weeks. Blood will be drawn at 0, 8, 12 and 52 weeks. Serum obtained from blood samples will be divided before being frozen at minus 20 degrees centigrade in each center. These serums will be transported to 'Hub' centers (to be selected), where they will be stored long-term; they shall not be transferred to any other party. These samples will be used to serotype the serological markers gASCA, pANCA, ACCA, ALCA and AMCA (serology profile). .

All participating gastroenterologists have agreed on standardized treatment regimens to be employed where possible and standardized follow-up protocols. The regimens and protocols were defined at a meeting held in Porto in June 2005 and validated at the meeting held in Porto in March 2007 . Use of standardized regimens removes treatment variability as a possible bias or confounding factor during disease outcome analysis. Institution of a second treatment, due to relapse or to lack of response, will be registered using a standardized relapse/lack of response form .

In general, multivariate statistical analysis will be employed to search for significant correlations between inflammatory and serological parameters and disease outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 0-18
* New onset Crohn's disease
* Treatment naive
* Ileocolonoscopy +radiology

Exclusion Criteria:

* Prior Treatment

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: New onset pediatric Crohn's disease until and including age 18
Sampling Method: Non-Probability Sample
Enrollment: 348 (Actual)
Dates: Start 2008-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Wolfson Medical center, Holon, Israel